CLINICAL TRIAL: NCT06024070
Title: Effect of Rigid Tapping on Chronic Functional Ankle Instability in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Gomaa Mohamed Eid, physiotherapist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012/003958
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Ankle Inversion Sprain

STUDY DESIGN:
Intervention Model Description: pre post study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): this study group assessed by 3 functional tests (Figure of 8 hopping , single leg stance test and y balance test) pre and post receiving rigid ankle tapping
  Interventions: Other: Rigid Tape

INTERVENTIONS:
Other: Rigid Tape — The patient was rested in supine or long sitting position on a table Pre-wrap was applied to cover all the area before tapping Two strips used separately as anchors at the two ends of the pre-wrap. Two Longitudinal stirrup of tape were used from medial side of the superior anchor to lateral side of the same anchor.
  Two horizontal stirrup of tape were used from medial side of the distal anchor to lateral side of the same anchor to support the medial side of the foot.
  Figure-of-eight straps were utilized for the taping. Lateral heel lock was applied.The tape then proceeded from the lateral side of the foot, looping around the heel, and returning to the same starting point by crossing over the Achilles tendon from behind.
  Medial heel lock was applied, the tape application was similar to the lateral heel lock but was at the opposite direction.
  Superior and inferior anchors were applied to support all the previous strips

SUMMARY:
This study aims rigid tapping on chronic functional ankle instability in professional basketball players.

DETAILED DESCRIPTION:
Lateral ankle sprains (LASs) are common injuries in sports and physical activities, with up to 40% of individuals experiencing a first-time LAS developing chronic ankle instability (CAI). LASs predominantly affect the anterior talofibular ligament, and residual symptoms can persist in a significant percentage of patients. However, many individuals with ankle sprains do not seek professional treatment, leading to potential underestimation of the injury severity. CAI is characterized by recurrent episodes of ankle giving way, ongoing symptoms, reduced ankle range of motion, diminished self-reported function, and persistent ankle sprains beyond one year. It is attributed to both mechanical and functional instability, with factors such as proprioceptive deficits and mechanical insufficiencies contributing to the condition. Taping, particularly rigid taping, is commonly used by athletes to enhance joint stability and improve dynamic balance and functional performance. Rigid taping limits joint movement, improves joint position, and provides external support without compromising functional performance. Taping is especially prevalent in multidirectional sports like basketball, where ankle sprains are frequent. The use of tapes aims to restrict ankle movement, increase joint stability, and enhance proprioception without hindering athletic performance.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players with age range from 18-40 years old.
* Body mass index (BMI) range from 18-25 H/m2.
* Participants had episodes of subjective sensation of instability in the last six months.
* Participants have at least moderate ankle instability, defined as a score of <25 on the Cumberland Ankle Instability Tool (CAIT).

Exclusion Criteria:

* Participants had a history of surgery or fractures in the ankle joints.
* Participants had a neurological or vestibular disorder.
* Participants were unable to understand the nature of the protocol and test instructions.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Ankle Stability | 3 days
  measured by y balance test and single leg stance test
functional performance | 3 days
  measured by Figure of 8 hopping test

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Fa Abdel-Majeed, phd, Study Chair — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No